CLINICAL TRIAL: NCT04169217
Title: Mentored Prehabilitation for Patients Having Aortic Aneurysm Surgery: a Pilot Randomised Control Trial
Brief Title: POWER: PrehabilitatiOn Workshop and Mentored Exercise Programme in Patients Having Elective Aortic Aneurysm Repair
Acronym: POWER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 241950
Record Dates: First submitted 2019-09-03; First posted 2019-11-19 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Vascular Surgery
Keywords: Prehabilitation
MeSH Terms: interventions — Preoperative Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control arm (No Intervention): This arm will not be in the prehabilitation group- as is current standard practice
- Group 2 (Active Comparator): This arm will be subject to a one off prehabilitation workshop and provided with a prehab booklet
  Interventions: Behavioral: Prehabilitation
- Group 3- Mentored group (Experimental): This arm will be subject to a one off workshop and provided with a prehab booklet- and additional mentoring by means of 1. an educational app, 2. push notifications,3. weekly communication with physiotherapy team member.
  Interventions: Behavioral: Prehabilitation

INTERVENTIONS:
Behavioral: Prehabilitation — A combination of a one off workshop and mentored prehabilitation.
  Covid Pandemic amendment: The workshop was originally a group based face to face patient workshop. This intervention is now (since the first national lockdown in March 2020) a virtual workshop using a the Bluejeans platform.
  Arms: Group 2; Group 3- Mentored group

SUMMARY:
Protocol Short Title:

POWER Study - PrehabilitatiOn Workshop and mentored Exercise programme in patients having elective aortic aneurysm Repair

Population:

Patients scheduled for elective repair of aortic aneurysm at St. Thomas' Hospital

Screening and recruitment:

Eligible participants will be identified by the vascular team; during the weekly multi-disciplinary team meeting, or via the clinical nurse specialist from tertiary referrals.

Participant information leaflets will then be sent out to eligible patients 2 weeks before the outpatient appointment.

Recruitment will be carried out during surgical outpatient appointments. Written informed consent will be obtained and participants will be randomised into three groups.

This pilot study will help us to:

1. To assess feasibility of screening, recruitment and retention
2. To assess adherence to intervention and blinding.
3. To generate outcome data that may be used to power definitive clinical trials

Primary objective To determine the feasibility of delivery of a randomised control trial.

Secondary objective (s) To determine baseline outcome data that may be used to power a randomised control trial.

Number of Subjects/Patients A convenience sample of 15 patients per group is planned, with a total of 45 patients recruited. At GSTT 200-250 aortic aneurysm operations are performed annually. We aim to recruit 40% of those eligible and screened. This would equate to 4-6 recruited per month.

Trial Design Single-blinded, randomised, controlled pilot study.

Patients will be allocated into the following groups:

Control group:

- Current standard practice, no prehabilitation workshop.

Non-mentored group:

* Prehabilitation workshop with no further patient contact.
* Participants to be given a prehab 'pack' which includes advice and a diary card.

Mentored group:

* Prehabilitation workshop with addition of regular 'mentoring' for up to 8 weeks after the workshop.
* Participants to be given a prehab 'pack' which includes advice and a diary card.

Primary Endpoints:

1. Screening and recruitment
2. Retention, blinding and follow up procedures.
3. Adherence

Secondary Endpoints:

To determine baseline outcome data that may be used to power a randomised control trial by examining the following:

1. Composite of post-operative cardiac, respiratory and renal complications at 30 days
2. Mortality at 30 days following surgery.
3. Length of postoperative hospital stay
4. Quality of life (EQ-5DL)- post surgery.
5. Tests of activity and function

Main Inclusion Criteria

Inclusion:

Elective all aortic aneurysm repair (Willingness to return after 8 weeks for re-assessment of secondary measures) Note: *COVID PANDEMIC ADJUSTMENT: Since March 2020, 1st national lockdown. Participants are no longer required to attend the 8 week follow up in person. The Quality of life questionnaires are done over the telephone by the research practitioner. The functional assessments are now done when the participant is admitted for their surgery Participants must have an e mail address.

Exclusions:

Urgent or emergency repair Contraindications to exercise (doesn't apply for short term illness) Severe musculoskeletal disorders preventing exercise

DETAILED DESCRIPTION:
Introduction

Optimising fitness prior to surgery, known as prehabilitation, has the potential to reduce risk and improve post-operative outcomes by increasing functional capacity and physiological reserve. Prehabilitation strategies include educating patients with lifestyle modifications such as smoking cessation, nutrition, exercise and anxiety reduction. Deconditioning and sarcopenia has been shown to predict a higher cost amongst patients undergoing major abdominal surgery [1] and has been recently identified as an independent predictor of hospital length of stay [2], hence optimising functionality may prevent morbidity.

There is a growing need to improve outcomes in vascular surgery, yet few examples of vascular prehabilitation exist. The 2018 Get It Right First Time (GIRFT) report [3] states one of the key recommendations is to improve the use of prehabilitation and to make it more consistent via NHS England commissioning.

Multiple studies with varying prehabilitation strategies have been published in the last decade [4]. Prehabilitation has been associated with encouraging results in major colorectal and upper gastrointestinal cancer surgery [5],[6]. Data such as these have also led to the development of prehabilitation services within NHS Trusts [7].

Supervised training programmes have shown to improve patient's anaerobic threshold and fitness in patients having aortic aneurysm repairs [8],[9],[10]. A recent randomised controlled trial has provided evidence to support supervised exercise training, by suggesting improvements in postoperative outcome, length of stay, postoperative pain and complications[11]. Historically there were concerns about exercising in this cohort of patients, however recent studies has shown that aneurysm expansion does not occur with exercise and exercise is safe [11],[12].

St. Thomas' Hospital is a tertiary referral centre performing between 200-250 aortic aneurysm repair operations annually. We serve a large demographic from South East England and receive referrals from across the whole of the UK, making the provision and appeal of a supervised prehabilitation exercise programme difficult.

Prehabilitation education provided is especially effective if delivered at the right time, for example, the need for high risk surgery; the so called 'teachable moment' [13]. Despite the recent surge in evidence surrounding the benefits of prehabilitation, it is not yet part of established pathways. There has been some guidance as to how to practically achieve prehabilitation into our clinical practice but there is still work to be done in terms of integrating it into perioperative pathways [14].

A mentored prehabilitation programme that does not require supervised exercise is generalisable and feasible, but yet to show improvements in patient outcomes.

Over the last 12 months we have been delivering a group based prehabilitation and exercise workshop named 'Road to Recovery'. This is a physiotherapist and anaesthetist led prehabilitation workshop, targeted to provide valuable education and advice to patients and their families about their surgery, hospital stay and expectations for discharge, diet, lifestyle and exercise before their aneurysm surgery. The advice emphasises the importance of empowering patients to take control of their own health. The workshop is designed to educate patients and allay their fears and anxieties around hospital admission and surgery.

The physiotherapist then provides a detailed lecture on exercise and the relevance of strength in the recovery period. An interactive, group-based demonstration of various safe and approved practical exercises is then undertaken. Feedback from the patients has been positive.

As part of the study, in addition to the prehabilitation workshop, we also aim to examine the potential benefits of a mentored approach, by use of technology and communication.

Our patients often live long distances from the hospital, so frequent hospital visits and supervised exercise sessions are not plausible. Therefore, a mentored prehabilitation programme could be considered more practical and generalisable.

We hypothesize that a prehabilitation workshop, and continued patient engagement, has the potential benefit to improve both the physical and psychological wellbeing of patients awaiting aortic aneurysm repair.

*COVID PANDEMIC ADJUSTMENT: Since March 2020, 1st national lockdown- We have made the workshops virtual rather than face to face. The participants and sent a link to join a virtual workshop, via the Bluejeans platform.*

An initial pilot study examining the study design and deliverability of a mentored approach prehabilitation programme, is warranted.

References

1. F. Gani et al., "Sarcopenia predicts costs among patients undergoing major abdominal operations," Surg. (United States), vol. 160, no. 5, pp. 1162-1171, 2016.
2. N. Shah et al., "The association of abdominal muscle with outcomes after scheduled abdominal aortic aneurysm repair," Anaesthesia, vol. 72, no. 9, pp. 1107-1111, 2017.
3. B. J. Orandi and J. H. Black, "Vascular Surgery," Curr. Surg. Ther., no. March, pp. 777-980, 2013.
4. K. Valkenet, I. G. van de Port, J. J. Dronkers, W. R. de Vries, E. Lindeman, and F. J. Backx, "The effects of preoperative exercise therapy on postoperative outcome: a systematic review," Clin. Rehabil., vol. 25, no. 2, pp. 99-111, 2011.
5. C. Li et al., "Impact of a trimodal prehabilitation program on functional recovery after colorectal cancer surgery: a pilot study and Other Interventional Techniques," Surg Endosc, vol. 27, pp. 1072-1082, 2013.
6. B. P. Chen et al., "Four-week prehabilitation program is sufficient to modify exercise behaviors and improve preoperative functional walking capacity in patients with colorectal cancer," Support. Care Cancer.
7. "Imperial College Healthcare | PREPARE programme." [Online]. Available: https://www.imperial.nhs.uk/our-services/cancer-services/oesophago-gastric-cancer/prepare-programme. [Accessed: 06-Sep-2018].
8. E. Kothmann et al., "Effect of short-term exercise training on aerobic fitness in patients with abdominal aortic aneurysms: A pilot study," Br. J. Anaesth., vol. 103, no. 4, pp. 505-510, 2009.
9. S. Pouwels, E. M. Willigendael, M. R. van Sambeek, S. W. Nienhuijs, P. W. Cuypers, and J. A. Teijink, "Beneficial Effects of Pre-operative Exercise Therapy in Patients with an Abdominal Aortic Aneurysm: A Systematic Review," Eur J Vasc Endovasc Surg, vol. 49, no. 1, pp. 66-76, 2015.
10. G. A. Tew et al., "Randomized feasibility trial of high-intensity interval training before elective abdominal aortic aneurysm repair," Br. J. Surg., vol. 104, no. 13, pp. 1791-1801, 2017.
11. H. M. Barakat, Y. Shahin, J. A. Khan, P. T. Mccollum, and I. C. Chetter, "Preoperative supervised exercise improves outcomes after elective abdominal aortic aneurysm repair," Ann. Surg., vol. 264, no. 1, pp. 47-53, 2016.
12. J. Myers et al., "A randomized trial of exercise training in abdominal aortic aneurysm disease," Med. Sci. Sports Exerc., vol. 46, no. 1, pp. 2-9, 2014.
13. P. Banugo and D. Amoako, "Prehabilitation," BJA Educ., vol. 17, no. 12, pp. 401-405, 2017.
14. G. A. Tew, R. Ayyash, J. Durrand, and G. R. Danjoux, "Clinical guideline and recommendations on pre-operative exercise training in patients awaiting major non-cardiac surgery," Anaesthesia, vol. 73, no. 6, pp. 750-768, 2018.

Our hypothesis is that a mentored prehabilitation programme will benefit patients having elective aortic aneurysm surgery. This approach should be tested in a pilot study to ensure appropriate study design, processes and uptake of the programme by patients.

Primary objectives

To determine the feasibility of delivery of a randomised controlled trial by examining the following:

1. Feasibility of screening and recruitment. Definition: screening: recruitment ratio of 3:1
2. Subject retention and adherence to 8-week follow up and blinding

Definition:

* Subject wearing activity tracker for greater than 80% of the time.
* 80% or more attendance to 8-week follow up.

  *COVID PANDEMIC ADJUSTMENT: Since March 2020, 1st national lockdown. Participants are no longer required to attend the 8 week follow up in person. The Quality of life questionnaires are done over the telephone by the research practitioner. The functional assessments are now done when the participant is admitted for their surgery
* 80% or more maintenance of blinding

  3. Adherence to trial protocol by comparing weekly physical activity between the three trial groups.
* Definition: increase in activity in intervention groups of 30% or more compared to the control group

Secondary objectives

To determine baseline outcome data that may be used to power a full randomised control trial by examining the following:

1. Composite of post-operative cardiac, respiratory and renal complications at 30 days

   Defined as:

   Cardiac: MI, new onset arrhythmia, prolonged inotropic support ( > 12 hours post op) Renal: renal insufficiency needing haemofiltration, >20% increase in creatinine from baseline.

   Respiratory: prolonged intubation > 12 hours, patient needing re- intubation, post-operative pneumonia
2. Mortality at 30 days
3. Length of hospital stay
4. Quality of life (QoL) EQ-5D-baseline, pre-operative, 6 weeks post-operative
5. Tests of activity and function using the following assessment tools at baseline and pre-operatively:

   * Duke Activity Status Index (DASI) score.
   * Time up and Go (TUAG)
   * Gait speed
   * Leg muscle strength

   Study Design This will be a single centre, single blinded, randomised, controlled pilot study.

   Inclusion criteria

   • Scheduled for aortic aneurysm surgery
   * Ability to walk
   * Willingness to wear the activity tracker for 8 weeks.
   * Willingness to return at 8 weeks for assessment of secondary outcomes

   Exclusion criteria
   * Urgent or emergency aneurysm repair
   * Patients who undergo emergency admission during the 8-week time frame, will be removed from the ongoing trial, but their data will be used up to that point.
   * Contraindications to exercise
   * Severe musculoskeletal disorders preventing exercise

   Recruitment

   Eligible patients will be identified either from tertiary referrals, or during the weekly aneurysm multidisciplinary meeting by the aortic clinical nurse specialist (CNS).

   The CNS will post the participant information leaflets to eligible participants 2-3 weeks before their first surgical consultation.

   The research team will then recruit and consent the participants on the day of their attendance to the surgical clinic.

   The workshop will run on two Fridays a month. The participants will then be randomised to one of three groups on this date. All recruited participants will be given the activity monitor and instructed on its use for the study.

   The participants recruited into the non-mentored (Arm 2) and mentored (Arm 3) interventions will then attend the workshop on the next available day. Participants in arm 3 will be given training on the use of the app.

   Participants will be reimbursed for all study-related travel costs.

   Randomisation

   Recruited participants will be randomised into one of three intervention groups in a 1:1:1 allocation ratio. A block randomisation technique with computer-generated sequence of random numbers will be produced using Sealed Envelope software (www.sealedenvelope.com).

   Study Arm 1 (Control):
   * Current usual practice, no prehabilitation workshop.

   Study Arm 2 (non-mentored prehabilitation):
   * Prehabilitation workshop with no further patient contact.
   * Participants to be given a prehab 'pack' which includes lifestyle advice.

   Study Arm 3 (mentored prehabilitation):
   * Prehabilitation workshop with regular 'mentoring' up to 8 weeks after the workshop, prior to their surgery.
   * Participants to be given a prehab 'pack' which includes lifestyle advice.
   * Weekly phone call by a member of the research team to remind and encourage the participant to increase activity.
   * Participants will be given a smartphone with a 'Prehab Activity' app. This app is designed and delivered by Medopad (London, UK). The app will include motivational push notifications, embedded documents and video clips summarising the importance of prehabilitation and demonstration of exercises.
   * The participants in this group will receive training in how to use the app by the research team.
   * Participants will have the opportunity to access expert advice from a designated physiotherapist in normal working hours.

   Medopad is a software company which provides health information and a learning platform for patients. All data is anonymised and the clinicians will be able to view any comments made by the participants (using their ID only) - this will be cleared once the participant finishes the trial.

   Medopad will receive anonymised feedback from participants via the research team.

   Activity Trackers All patients are to have their activity levels tracked by an Actiwatch Spectrum (PHILIPS Healthcare, Eindhoven, Netherlands) activity tracker. This is a lightweight, waterproof, wrist-worn device. All data will be stored on the trackers and downloaded anonymously onto secure research computers for analysis.

   Outcome assessors will be blinded to the intervention.

   Follow up

   Patients will be followed at two time points in the trial, prior to surgery after the eight-week intervention period (Follow up 1) and six weeks post-operatively (Follow up 2).

   Follow up 1: Eight weeks after recruitment, prior to surgery

   - The participant will be requested to attend St Thomas' Hospital to complete a QoL questionnaire and functional assessments.

   NOTE: *COVID PANDEMIC ADJUSTMENT: Since March 2020, 1st national lockdown. Participants are no longer required to attend the 8 week follow up in person. The Quality of life questionnaires are done over the telephone by the research practitioner. The functional assessments are now done when the participant is admitted for their surgery , which is not necessarily at 8 weeks.

   - The outcome assessor will remain blinded to the group allocation of the participant.

   Follow up 2: Six weeks postoperative Subjects will be contacted to complete a QoL questionnaire. Electronic patient records and discharge letters will be used to collect data on post-operative complications, 30-day mortality and length of hospital stay.

   Data Recording All data will be recorded onto paper CRFs which will then be transferred onto CASTOR database.

   Data collection

   Demographics Co-morbidities Size and type of aneurysm Surgical method

   Baseline data: Day 1; Surgical Consultation Co-morbidities Renal function QoL: EQ-5D

   Functional assessment:
   * Duke Activity Status Index Score
   * Gait speed
   * 'Timed up and Go'
   * Hip flexion strength

     8 weeks: After the surgical OPA, before surgery. Repeat of the functional assessments and QoL assessment.

   Postoperative data:

   - Composite of post-operative cardiac, respiratory and renal complications at 30 days
   * Death at 30 days
   * Length of hospital stay
   * EQ-5D

ELIGIBILITY:
Inclusion Criteria:

* • Attending GSTT for aortic aneurysm surgery

  * Ability to walk (determined by ability to perform gait speed independently)
  * Willingness to wear the activity tracker for 8 weeks.
  * Willingness to return at 8 weeks for re-assessment of secondary outcome measures: Note: *COVID PANDEMIC ADJUSTMENT: Since March 2020, 1st national lockdown.

Participants are no longer required to attend the 8 week follow up in person. The Quality of life questionnaires are done over the telephone by the research practitioner. The functional assessments are now done when the participant is admitted for their surgery

Exclusion Criteria:

* Urgent or emergency aneurysm repair

  * Patients who undergo emergency admission during the 8-week time frame, will be removed from the ongoing trial, but their data will be used up to that point.
  * Contraindications to exercise (doesn't apply for short term illness ( appendix 4).
  * Severe musculoskeletal disorders preventing exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-02-02 (Actual)

PRIMARY OUTCOMES:
Feasibility of screening and recruitment: recruitment ratio | 18 months
  Screening: recruitment ratio of 3:1
Subject retention and adherence to 8-week follow up and blinding | 8 weeks
  Subject wearing activity tracker for greater than 80% of the time, 80% or more attendance to 8-week follow up * and 80% or more maintenance of blinding.
  *COVID PANDEMIC ADJUSTMENT: Participants are no longer required to attend the 8 week follow up in person. The Quality of life questionnaires are done over the telephone by the research practitioner. The functional assessments are now done when the participant is admitted for their surgery
Adherence to trial protocol by comparing weekly physical activity between the three trial groups. | 18 months
  Increase in activity in intervention groups of 30% or more compared to the control group as measured by the actiwatch

SECONDARY OUTCOMES:
Composite of post-operative cardiac complications at 30 days | 30 days post surgery.
  MI, new onset arrhythmia, prolonged inotropic support ( > 12 hours post op)
Composite of post-operative respiratory complications at 30 days | 30 days post surgery
  Prolonged intubation > 12 hours, patient needing re- intubation, post-operative pneumonia
Composite of post-operative renal complications at 30 days | 30 days post surgery
  renal insufficiency needing haemofiltration, >20% increase in creatinine from baseline.
Mortality at 30 days | 30 days post surgery
  Mortality status of those in each group at 30 days
Length of hospital stay | 18 months
  How long each participant in each group stayed in hospital post surgical intervention
Quality of life (QoL) EQ-5D | 18 months
  Participants QoL through the study - baseline, pre-operative and 6 weeks post-operative. This may be unto 18 months.
Tests of activity and function | 8 weeks
  Duke Activity Status Index (DASI) score at baseline and at 8 weeks
Tests of activity and function | 8 weeks
  'Timed up and Go'- at baseline and 8 weeks
Tests of activity and function | 8 weeks
  Gait speed- at baseline and 8 weeks
Tests of activity and function | 8 weeks
  Leg Strength measured by hand held dynamometer- at baseline and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Heena Bidd, Study Chair — Guys & St Thomas' NHS Foundation Trust
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bidd H, Wong DJN, Colville G, Banugo P, Baldwin M, Waring H, Zucco L, Radcliife G, Zayed H, El-Boghdadly K. Mentored multimodal prehabilitation for aortic aneurysm surgery: a pilot randomised controlled trial. Perioper Med (Lond). 2025 Nov 22;14(1):132. doi: 10.1186/s13741-025-00625-6. PMID 41275253